CLINICAL TRIAL: NCT07053995
Title: EFFECTIVENESS OF PREOPERATIVE VAGINAL CLEANING IN REDUCING POST CAESAREAN INFECTIOUS MORBIDITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Naba Rehman, Consultant, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 978
Record Dates: First submitted 2025-06-23; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Endometrial; Infection; Surgical Site Infection Following Cesarean Delivery
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with vaginal cleaning (Experimental): Total of 38 participants included randomly after informed consent. Vaginal cleaning with 50cc (0.5cc chlorhexidine) along with abdominal scrubbing was done before giving incision for C-section. Prophylactic antibiotics were given. Participants were followed and incision site was inspected on day 14. Data was recorded.
  Interventions: Procedure: Vaginal cleaning
- Participants with non vaginal cleansing (Other): Total of 38 participants included randomly after informed consent. Only routine abdominal scrubbing was done before giving incision for C-section. Prophylactic antibiotics were given. Participants were followed and incision site was inspected on day 14. Data was recorded.
  Interventions: Other: Non vaginal cleansing

INTERVENTIONS:
Procedure: Vaginal cleaning — Before giving incision for C-section surgery, vaginal cleaning was done with 50cc diluted antiseptic solution as a single push.
  Arms: Participants with vaginal cleaning
Other: Non vaginal cleansing — Routine abdominal scrubbing was carried out before incision. No vaginal cleaning was done before incision.
  Arms: Participants with non vaginal cleansing

SUMMARY:
After obtaining an informed consent a detailed history and clinical examination was performed. Labs were carried out to fulfill inclusion and exclusion criteria. Women were randomly divided into two groups. In Intervention group vaginal cleaning was done with 50cc diluted antiseptic solution where as control group had abdominal scrub only. Participants were followed and incision site was checked at day 14.

DETAILED DESCRIPTION:
After obtaining an informed consent a detailed history and clinical examination was performed. Labs were carried out to fulfill inclusion and exclusion criteria. Women were randomly divided into two groups. In Intervention group vaginal cleaning was done with 50cc diluted antiseptic solution as single push where as control group had abdominal scrub only. Participants were followed and incision site was checked at day 14. Data was recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 18-40 years
* Gestational age greater than 36 weeks undergoing elective C section

Exclusion Criteria:

* Pregnant women with history of allergic reactions to chlorhexidine
* Placenta previa on ultrasound scan
* Diabetes Mellitus on fasting blood sugar
* Anemia (Hb less than 7g/dl)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Endometrial Infection | 14 days
  Body temperature was measured postoperatively along with any dicharge of pain around uterine region 24hrs after surgery
Surgical site infection | 14 days
  Incision site was inspected on 4th and 14th post operative day and documented any evidence of infection signs according to Southampton wound grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hira Hassan, MBBS FCPS, Study Director — Khyber Teaching Hospital Peshawar
Locations (1):
- Khyber Teaching Hospital Peshawar Pakistan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No